CLINICAL TRIAL: NCT02668796
Title: A Phase III Investigator-Blind, Randomized, Parallel-Group, Placebo- Controlled, Multicentre Study to Evaluate the Therapeutic Equivalence and Safety of Estradiol Vaginal Tablets 10 mcg and Vagifem® (Estradiol Vaginal Tablets) 10 mcg (Novo Nordisk Inc.) Administered for 14 Days and Compare Both Active Treatments to a Placebo Control in Female Subjects With Moderate to Severe Symptoms of Vulvar and Vaginal Atrophy Associated With Menopause.
Brief Title: To Study Generic Estradiol 10 mcg Vaginal Tablets in the Treatment of Vulvar and Vaginal Atrophy in Post Menopausal Women.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLK-1502
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2016-09

CONDITIONS: Vulvar and Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol Vaginal Tablets 10 mcg (Glenmark) (Experimental): apply using the given applicator
  Interventions: Drug: Estradiol Vaginal Tablets 10 mcg (Glenmark)
- Vagifem® (Estradiol Vaginal Tablets) 10 mcg (Novo Nordisk) (Active Comparator): apply using the given applicator
  Interventions: Drug: Vagifem® (Estradiol Vaginal Tablets) 10 mcg (Novo Nordisk)
- Placebo of Estradiol Vaginal Tablets 10 mcg (Glenmark) (Placebo Comparator): apply using the given applicator
  Interventions: Drug: Placebo of Estradiol Vaginal Tablets 10 mcg (Glenmark)

INTERVENTIONS:
Drug: Estradiol Vaginal Tablets 10 mcg (Glenmark) — apply using the given applicator
  Arms: Estradiol Vaginal Tablets 10 mcg (Glenmark)
Drug: Vagifem® (Estradiol Vaginal Tablets) 10 mcg (Novo Nordisk) — apply using the given applicator
  Arms: Vagifem® (Estradiol Vaginal Tablets) 10 mcg (Novo Nordisk)
Drug: Placebo of Estradiol Vaginal Tablets 10 mcg (Glenmark) — apply using the given applicator
  Arms: Placebo of Estradiol Vaginal Tablets 10 mcg (Glenmark)

SUMMARY:
This is a Randomized, Parallel-Group, Placebo- Controlled, Multicenter Study to Evaluate the Therapeutic Equivalence and Safety of Estradiol Vaginal Tablets 10 mcg and Vagifem® (Estradiol Vaginal Tablets) 10 mcg (Novo Nordisk Inc.) in Female Subjects with Moderate to Severe Symptoms of Vulvar and Vaginal Atrophy Associated with Menopause.

ELIGIBILITY:
Inclusion Criteria:

1. Female postmenopausal subjects aged >30 to <75 years
2. At least 1 subject assessed moderate to severe symptom of vulvar and vaginal atrophy among the following that is identified as being the most bothersome to her

   * vaginal dryness
   * vaginal and/or vulvar irritation/ itching
   * dysuria
   * vaginal pain associated with sexual activity
   * presence of vaginal bleeding associated with sexual activity
3. Have <5% superficial cells on vaginal smear cytology and vaginal pH >5.0 at Visit 1
4. Systolic blood pressure <150mm Hg and diastolic blood pressure <90mm Hg at Visit 1

Exclusion Criteria:

1. Known hypersensitivity to Estradiol vaginal tablet
2. Screening mammogram or clinical breast examination results indicating any suspicion of breast malignancy.
3. History of undiagnosed vaginal bleeding.
4. History of significant risk factors for endometrial cancer
5. For women with an intact uterus, screening vaginal ultrasonography showing endometrial thickness of ≥ 4 mm.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with at least 25% reduction from baseline in the sum of % basal/parabasal + %intermediate cells on vaginal cytology and vaginal pH <5.0 with a change from baseline vaginal pH of at least 0.5 | Day 15]

SECONDARY OUTCOMES:
The proportion of subjects with treatment success at the end of study where treatment success is defined as a subject who achieves a score of 0 (none) or 1 (mild) at Visit 3/End of Study for the MBS | Day 15]

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nikhil Sawant, Study Director — Glenmark Pharmaceuticals Ltd.
Locations (1):
- Glenmark Pharmaceuticals Inc., Mahwah, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No